CLINICAL TRIAL: NCT00351715
Title: Sublingual Methadone for the Management of Cancer-related Breakthrough Pain in Outpatients: a Phase II Multicenter, Open Label, Feasibility Study
Brief Title: Sublingual Methadone for the Management of Cancer-related Breakthrough Pain in Outpatients
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study stopped due to low accrual
Sponsor: AHS Cancer Control Alberta (Other)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20144; 22206
Record Dates: First submitted 2006-07-11; First posted 2006-07-13 (Estimated); Last update posted 2019-10-21 (Actual); Status verified 2008-10

CONDITIONS: Cancer; Pain
Keywords: Sublingual Methadone; Cancer related breakthrough pain; feasibility study; Phase II/open label; Outpatients; Safety/ efficacy; previously receiving opioids; speak English
MeSH Terms: conditions — Neoplasms; Pain

ARMS (1):
- Pharmacokinetic (Experimental): One episode of breakthrough pain was to be evaluated per patient. Clinical status and bloodwork was evaluated prior to entering into this phase of the trial, and patients were eligible if bloodwork demonstrated a HgB of >90 g/L with no concurrent bleeding. A peripheral intravenous catheter was inserted and saline locked. When breakthrough pain was experienced, methadone was administered, and the patient completed a pain intensity numeric rating scale at time 0 and every 10 minutes for one hour. A 10 cc specimen of blood was collected prior to administration of methadone, and again every 10 minutes for one hour. Blood was collected without anticoagulant, allowed to clot, separated by centrifugation, and serum samples flash frozen. Serum methadone levels were quantified by LC/MS/MS with comparison to isotopically labeled internal standards
  Interventions: Drug: Sublingual Methadone

INTERVENTIONS:
Drug: Sublingual Methadone

SUMMARY:
The purpose of this Phase II study is to determine the feasibility of the dose titration and assessment protocol in the outpatient population before conducting an appropriately powered phase III study. Thus the primary purpose of this study is to determine the proportion of patients who are successfully titrated to an optimal dose of sublingual (Under the tongue) methadone and then studied at that optimal dose with successive episodes of breakthrough pain.

ELIGIBILITY:
Inclusion Criteria:

* Pain due to cancer or its treatment; controlled baseline pain;
* episodes of breakthrough pain every day that are "4/10" in severity or greater, ;
* ast 10 minutes or longer, and
* are responsive to short acting oral opioids such as morphine or hydromorphone;
* are able to hole a volume of 1.0cc of water under the tongue for a 5-minute period; are able to provide written informed consent;
* are able to fill out the study forms

Exclusion Criteria:

* Severe underlying respiratory disease such that an investigator is wary about the risk of respiratory failure from modest doses of opioid;
* prior sensitivity to methadone;
* currently are being administered methadone;
* have breakthrough pain that in the opinion of the investigator is likely to change within the next seven days (recent or imminent radiation therapy to the main site of pain,
* new chemotherapy or use of an injectable bisphosphonate likely to alter the pain, new use corticosteroids within the past week with a corresponding change in pain, or other interventions judged likely to alter pain);
* are clinically unstable or have a life expectancy of less than one month making completion of the trial unlikely

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2008-07; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

PRIMARY OUTCOMES:
to demonstrate the feasibility of a novel model to assess sublingual methadone to breakthrough pain in the outpatient setting | 12 months

SECONDARY OUTCOMES:
to develop a model of PK/PD study of breakthrough pain | Baseline to 5 years
to develop a research tool, the Breakthrough Pain Assessment Tool (BPAT) | Baseline to 5 years
to demonstrate proof of concept | Baseline to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Neil Hagen, MD, Principal Investigator — AHS Cancer Control Alberta
Locations (2):
- Canada (2):
  - Tom Baker Cancer Center, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta